CLINICAL TRIAL: NCT00002621
Title: A Phase II Study of Alpha Interferon (alphaIFN) In HIV-Related Malignancies - A Pediatric Oncology Group Wide Study
Brief Title: Interferon Alfa in Treating Children With HIV-Related Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9362; POG-9362 (Other: Pediatric Oncology Group); CDR0000063972 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2003-08-11 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Leukemia; Lymphoma; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: recurrent childhood acute lymphoblastic leukemia; stage I childhood lymphoblastic lymphoma; stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; unspecified childhood solid tumor, protocol specific; untreated childhood acute myeloid leukemia and other myeloid malignancies; untreated childhood acute lymphoblastic leukemia; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; stage I childhood small noncleaved cell lymphoma; stage I childhood large cell lymphoma; stage II childhood small noncleaved cell lymphoma; stage II childhood large cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood small noncleaved cell lymphoma; stage IV childhood large cell lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating | interventions — Interferon-alpha; Introns; Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alpha interferon (aIFN) treatment (Experimental): See detailed description.
  Interventions: Biological: recombinant interferon alfa

INTERVENTIONS:
Biological: recombinant interferon alfa
  Other Names: Intron A; Roferon A; NSC 377523

SUMMARY:
RATIONALE: Interferon alfa may interfere with the growth of cancer cells.

PURPOSE: Phase II trial to study the effectiveness of interferon alfa in treating children with an HIV-related cancer including leukemia, non-Hodgkin's lymphoma, CNS lymphoma, or other solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the complete response rate and one-year disease free survival of pediatric patients with HIV-related malignancies treated with interferon alfa.
* Determine the toxicity of interferon alfa alone and in combination with antiretroviral therapy in these patients.

OUTLINE:

* Induction: Patients receive interferon alfa subcutaneously (SC) daily on days 1-14. Patients with advanced stage III or IV undifferentiated lymphomas or B-cell acute lymphoblastic leukemia also receive hydrocortisone intrathecally (IT) combined with cytarabine IT on day 14.
* Maintenance: Patients with stable or responding disease after completion of induction receive interferon alfa SC 3 times a week beginning on week 1. Treatment continues for a minimum of 4-12 weeks in the absence of disease progression or unacceptable toxicity. Patients who received IT therapy during induction receive the same IT therapy at 4, 8, and 12 weeks and then every 8 weeks thereafter.

Patients are followed every 6 months for 4 years and then annually for survival until entry on another POG protocol.

PROJECTED ACCRUAL: A total of 14-30 evaluable patients will be accrued for this study within 4.2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven malignancy diagnosed at any time following confirmation of HIV-positivity, including the following:

  * Leukemia
  * Non-Hodgkin's lymphoma
  * CNS lymphoma
  * Other solid tumors
* Measurable disease
* Concurrent registration on protocol POG-9182 required

  * Confirmed HIV-positive by POG-9182 criteria
  * Required biology studies completed

PATIENT CHARACTERISTICS:

Age:

* 21 and under

Performance status:

* Not specified

Life expectancy:

* More than 4 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3 (unless bone marrow involvement present)

Hepatic:

* See Disease Characteristics
* Bilirubin less than 1.5 times normal
* SGPT and SGOT less than 2 times normal (may discuss with Study Coordinator)

Renal:

* Creatinine less than 1.5 mg/dL

Cardiovascular:

* Adequate cardiac function by echocardiogram/MUGA scan

Other:

* Chronically infected patients must be stable enough to meet life expectancy requirement

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior interferon for cancer
* Prior interferon alfa for viral infections (i.e., hepatitis) must be discussed with Study Coordinator

Chemotherapy:

* At least 1 week since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 1 week since prior radiotherapy

Surgery:

* Not specified

Other:

* Prior antiretroviral therapy allowed
* At least 1 week since prior acute treatment for any serious or life-threatening infection
* No concurrent local treatment unless discussed with the Study Coordinator
* No concurrent acute treatment for any serious or life-threatening infection
* Concurrent antiretroviral therapy allowed

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 1994-12; Primary Completion 2002-07 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Complete response rate for HIV related malignancies treated with interferon | Length of study

SECONDARY OUTCOMES:
Event Free Survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: V. M. Whitehead, MD, Study Chair — Montreal Children's Hospital at McGill University Health Center
Locations (10):
- United States (7):
  - Via Christi Regional Medical Center, Wichita, Kansas
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tomorrows Children's Institute, Hackensack, New Jersey
  - Mission Saint Joseph's Health System, Asheville, North Carolina
  - Medical City Dallas Hospital, Dallas, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
- McGill University Health Center - Montreal Children's Hospital, Montreal, Quebec, Canada
- University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan, Puerto Rico
- Clinique de Pediatrie, Geneva, Switzerland